CLINICAL TRIAL: NCT06393777
Title: Effectiveness of Pre-administered Natural Sweet-tasting Solution (Honey) for Decreasing Pain Associated With Dental Injections (Infiltration) Prior to Extraction in 6-8 Years Old Children In Comparison to Topical Anesthesia. (RCT)
Brief Title: Effectiveness of Pre-administered Natural Sweet-tasting Solution (Honey) for Decreasing Pain of Needle Insertion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Lotfy Mohamed Saleh, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pain of dental injection pedo
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Analgesia
Keywords: honey; injection; local anesthesia; pain
MeSH Terms: conditions — Agnosia; Pain | interventions — Honey

STUDY DESIGN:
Intervention Model Description: This trial is a randomized clinical trial (parallel design 1:1).
Who Masked: Participant, Outcomes Assessor
Masking Description: This research will be a double blinded study, where the patient (participant) and the statistician will be blind to the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Pre-administered honey for Decreasing Pain of Dental Injections (Experimental): The participants were asked to drink 5 mL of honey solution before injecting on the experimental side, the patient was asked to hold the solution in the mouth for a minute and then to spit it out .
  Interventions: Dietary Supplement: honey
- topical anesthesia (Other): benzocaine 20% gel was applied to the test sites on side of the jaw with a cotton tip applicator which was completely soaked for a period of 5 minutes.
  Interventions: Dietary Supplement: honey

INTERVENTIONS:
Dietary Supplement: honey — analgesic effect of honey

SUMMARY:
This study aims to assess Effectiveness of Pre-administered Natural Sweet-tasting Solution (honey) for Decreasing Pain Associated with Dental Injections (infiltration) prior to dental extraction in 6-8 years old healthy Children (first dental visit) In comparison to topical anesthesia.

DETAILED DESCRIPTION:
The administration of local anesthetics is one of the most dreaded or anxiety-inducing triggers in a dental setup. Patients, particularly children, may be fearful of dental injections, which may prevent them from seeking dental treatment. Even though profound local anesthesia aids in the treatment of pediatric patients in terms of reducing their anxiety and pain during restorative and surgical procedures, the fear of needles has been cited as a barrier to develop proper dental care. Numerous techniques have been researched in an attempt to minimize the pain and distress associated with these dental injections, varying from localized methods to distraction techniques. The localized methods include application of topical agents, altering the rate of injection, increasing the pH of local anesthetics by buffering and pretreatment with lasers. Instruments such as CCLA System (computer-controlled local anesthetic delivery system) and dental vibe are also available to make dental injections more comfortable. Studies have found that sweet flavored solutions, mainly 30% sucrose, given orally prior to cutaneous procedures can reduce discomfort in neonates undergoing heel sticks and venipuncture. Effectiveness of sucrose in the treatment of, procedural pain in newborns and babies has been verified in a Cochrane reviews.

ELIGIBILITY:
Inclusion Criteria:

1. Children within the age group 6 to 8 years were selected since the cognitive skills necessary for the use of visual analogue scale for pain assessment have not developed in children younger than 6 years of age.
2. Mobile deciduous second molars bilaterally that could be treated under infiltration anesthesia.

Exclusion Criteria

1. History of allergy to any components of local anesthetic agents used during the study.
2. Dental or dentoalveolar abscess.
3. Presence of any underlying systemic disease.
4. Immunocompromised patients.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain perception during Dental injection Dental injection Pain perception during Dental injection | 1 year
  Wong-Baker ratting scale 0 happy ,2 hurts a little bit,4 "hurts a little more"6 hurts even more,8 hurts a whole lot"10hurts worst" Rating scale Wong-Baker Rating scale

SECONDARY OUTCOMES:
Child behavior during dental injection | 1 year
  The SEM(sound, eye, motor) scale Scale from (0-4)

OTHER OUTCOMES:
heart rate during dental injection | through study completion, an average of 1 year".
  Pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan Omar Elgebaly, Lecturer, Principal Investigator — Outpatient clinic, department of Pediatric Dentistry, Faculty of Dentistry, Cairo University.

REFERENCES:
- [Background] Janiani P, Gurunathan D. Effectiveness of Pre-administered Natural Sweet-tasting Solution for Decreasing Pain Associated with Dental Injections in Children: A Split-mouth Randomized Controlled Trial. J Contemp Dent Pract. 2021 Dec 1;22(12):1434-1437. PMID 35656683
- [Background] Gumus H, Aydinbelge M. Evaluation of effect of warm local anesthetics on pain perception during dental injections in children: a split-mouth randomized clinical trial. Clin Oral Investig. 2020 Jul;24(7):2315-2319. doi: 10.1007/s00784-019-03086-6. Epub 2019 Oct 24. PMID 31650314